CLINICAL TRIAL: NCT02825914
Title: CAsein GLycomacropeptide in Ulcerative Colitis - Anti-Inflammatory and Microbiome Modulating Effects (CAGLUCIM)
Acronym: CAGLUCIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAGLUCIM2016
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Colitis, Ulcerative; Inflammatory Bowel Diseases
Keywords: glycopeptides; human microbiome; caseinomacropeptide; whey protein; dietary proteins
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Casein glycomacropeptide (CGMP) (Active Comparator): As add-on to the standard medical treatment of active ulcerative colitis the patients will receive a daily oral intake of CGMP-protein-shake during 12 weeks.
  Interventions: Dietary Supplement: Casein glycomacropeptide (CGMP)
- Placebo (Placebo Comparator): As add-on to the standard medical treatment of active ulcerative colitis the patients will receive a daily oral intake of placebo-shake consisting of milk powder during 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Casein glycomacropeptide (CGMP)
  Arms: Casein glycomacropeptide (CGMP)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Casein glycomacropeptide (CGMP) has anti-inflammatory properties in experimental rodent colitis and using human in vitro inflammation models. Its use as a food ingredient has proven safe and with no influence on dietary intake. In a pilot study the investigators found, that orally administered CGMP seems to have a beneficial effect comparable to that of mesalazine in active distal ulcerative colitis.

The investigators wish to evaluate the effects in a larger group of patients with active ulcerative colitis by studying the clinical effects and assessing the anti-inflammatory and microbiome modulating properties.

ELIGIBILITY:
Inclusion Criteria:

* ulcerative colitis (verified by mucosal histology and endoscopy)
* Clinically active ulcerative colitis (SCCAI ≥ 3)

Exclusion Criteria:

* Endoscopically inactive disease (Endoscopic Mayo Score of 0)
* Lactose or milk protein intolerance
* Celiac disease
* Not able to understand or speak Danish.
* Pregnant or nursing.
* Growth of pathogenic bacteria in stool culture from 4 weeks before and until randomization (Salmonella, Campylobacter, Yersinia or Clostridium Difficile.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Endoscopic remission | 12 weeks
  The number of patients in endoscopic remission/macroscopic mucosal healing (Endoscopic Mayo Score of 0)
Clinical remission | 12 weeks
  The number of patients in clinical remission (SCCAI ≤ 2)
Clinical Response | 12 weeks
  The number of patients with clinical response (reduction of SCCAI-score of at least 2 points)
Fecal inflammatory marker | 12 weeks
  The number of patients with a fecal-calprotectin below 150 mg/kg

SECONDARY OUTCOMES:
Endoscopic response | 12 weeks
  The number of patients with endoscopic response (reduction of Endoscopic Mayo Score of at least 1point)
Steroid-free remission | 12 weeks
  The number of patients in steroid-free remission (SCCAI ≤ 2)
Clinical remission at follow-up | 26 weeks
  The number of patients in clinical remission (SCCAI ≤ 2)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik A Vilstrup, Professor, Study Chair — University of Aarhus
Locations (1):
- Department of medicine V (Hepatology and Gastroenterology), Aarhus C, Denmark